CLINICAL TRIAL: NCT04509908
Title: Eating and Physical Activity Patterns of the Population Working in the Uruguayan State Electrical Company.
Acronym: PAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Administración Nacional de Usinas y Transmisiones Eléctricas (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government); Universidad de la Republica (Other); Universidad de Granada (Other)
Responsible Party: Principal Investigator, Mercedes Medina Vadora, EATING AND PHYSICAL ACTIVITY PATTERNS OF THE POPULATION WORKING IN THE URUGUAYAN STATE ELECTRICAL COMPANY., Administración Nacional de Usinas y Transmisiones Eléctricas
Other Study IDs: MMVadora
Record Dates: First submitted 2020-07-23; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Diet Habit; Weight, Body
Keywords: Diet; Work related; physical activity
MeSH Terms: conditions — Feeding Behavior; Body Weight; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stuydy of eatin and physical activity patterns in Uruguayan workers and association with obesity, overweight, and tasks.

DETAILED DESCRIPTION:
A sample of workers from the electrical company will be studies as to eating and physical activity patterns, weight variations, and assigned tasks.

ELIGIBILITY:
Inclusion Criteria:

* It will include all the officials who joined the company from January 1, 2010 to December 31, 2017, of whom they are between 18 and 65 years old, and the total was from 1964.

Exclusion Criteria:

* On the other hand, regarding the officials who meet the inclusion criteria, the following exclusion criteria are established. Therefore, those officials who:

  * Do not have a medical check-up at admission and at least one checkup between one year and two years after entering the company
  * Officials who no longer continue to work at the institution at the date of the study.
  * Participants who do not have weight and height recorded in the medical record

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It will include all the officials who joined the company from January 1, 2010 to December 31, 2017. They are 1964 aged between 18 and 65 years old.They are living in Montevideo and 416 are women and 1,548 are men.
Sampling Method: Non-Probability Sample
Enrollment: 1964 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Weight | 2010 at 2020
  weight in kilograms will be taken records and in person from 2010
Height | 2010 at 2020
  Height in meters will be taken records and in person from 2010
Body mass index | 2010 at 2020
  body mass index in weight / meters squared

SECONDARY OUTCOMES:
Diet by 24 hours recall | 2020
  Diet in investigated with 24 hours recall
Diet by frequency of food consumption | 2020
  Frequency of food consumption semi-qualitative

OTHER OUTCOMES:
Physical activity | 2020
  Physical activity will be measured with International Physical Activity Questionnaires (IPAQ)
Acelerometer | 2020
  The accelerometer is shown as one of the most accurate techniques in recording and saving the amount and level of physical activity, by each person in a given period of time.
Typs of job | 2010 at 2020
  sedentary or active type of work

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Lecot, Dr., Principal Investigator — Servicio Medico UTE - Sta Fe 1041, 11800 Montevideo, Uruguay
Locations (1):
- Servicio Medico - UTE, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Medina-Vadora MM, Severi C, Lecot C, Ruiz-Lopez MD, Gil A. Study of Food Intake and Physical Activity Patterns in the Working Population of the Uruguayan State Electrical Company (UTE): Design, Protocol and Methodology. Nutrients. 2021 Oct 9;13(10):3545. doi: 10.3390/nu13103545. PMID 34684546